CLINICAL TRIAL: NCT01593605
Title: Resveratrol-Leucine Metabolite Synergy in Pre-diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Nutraceutical Discoveries, Inc. (Other)
Responsible Party: Principal Investigator, Wanda Snead, Study Sub-Investigator/Coordinator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KNIS-NCI
Record Dates: First submitted 2012-05-02; First posted 2012-05-08 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Impaired Glucose Tolerance
Keywords: Impaired glucose tolerance, pre-diabetes,glycemic control,; supplements
MeSH Terms: conditions — Glucose Intolerance | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dietary Supplement/insulin sensitivity (Active Comparator): The first study supplement contains resveratrol that may improve insulin sensitivity and Leucine.Resveratrol 50mg with leucine 1.11 g. - one tablet taken twice a day by mouth
  Interventions: Dietary Supplement: Resveratrol
- Sugar Pill (Placebo Comparator): Neutral treatment Placebo - one tablet taken twice a day by mouth
  Interventions: Other: Placebo treatment
- Dietary Supplement 2 (Active Comparator): 2nd study supplement contains resveratrol and HMB which may stimulate protein building.
  Interventions: Dietary Supplement: resveratrol /HMB

INTERVENTIONS:
Dietary Supplement: Resveratrol — A blend of low dose resveratrol and either leucine or HMB will be useful nutraceutical strategies for the control of elevated blood glucose in non-diabetic individuals with elevated fasting glucose. The proposed project is designed to evaluate this hypothesis by comparing the effects of resveratrol (50 mg)/leucine (1.11 g) administered twice daily (bid).
  Arms: Dietary Supplement/insulin sensitivity
Dietary Supplement: resveratrol /HMB — resveratrol (50 mg)/HMB (500 mg) twice daily (bid) with placebo on fasting blood glucose, glucose tolerance, insulin, C-peptide, glucagon, fructosamine and F2-isoprostanes in non-diabetic subjects with elevated fasting blood glucose.
  Arms: Dietary Supplement 2
Other: Placebo treatment — Placebo - one tablet taken twice a day by mouth
  Arms: Sugar Pill

SUMMARY:
The study will evaluate the effects of resveratrol/leucine and resveratrol/HMB for their ability to control glucose levels in persons without diabetes but with impaired fasting glucose. Secondary assessments will examine the effect of these nutritional supplements versus placebo on inflammation, fasting lipids, HbA1C, and fructosamine, longer term metabolic markers of risk in diabetes.

DETAILED DESCRIPTION:
This will be a 28-day randomized controlled trial of the effects of a nutraceutical preparation on glycemic control in non-diabetic individuals with impaired glucose tolerance (IGT). IGT will be defined by American Diabetes Association criteria, as outlined in the list of inclusion and exclusion criteria (copy attached). There will be two active treatment arms and a placebo arm (3 arms total, n=12 completed subjects per arm). Following screening for inclusion/exclusion criteria and obtaining informed consent, subjects will be enrolled in the study and provided instructions to maintain their usual dietary pattern and physical activity level. If recent physical examination and medical history are not available; H&P will be conducted and recorded for each enrolled subject. Subjects will be instructed to follow a 12-hour fast starting on day -1, and on the morning of day 0 fasting blood is drawn for analyses indicated below and the supplements are distributed. Supplements are distributed using a blinding protocol and a variable, known pill allotment in order to assess compliance via standard pill counts. Pill bottles and all unused supplements are returned at seven day intervals, with new supplies being distributed at that time. Fasting blood samples are obtained on days 0, 7, 14 and 28. Samples from each day are analyzed for glucose and insulin. Samples from days 0, 14 and 28 are also analyzed for fructosamine, C-peptide, glucagon and F2-isoprostanes. A75 g oral glucose tolerance test administered on days 0 and 28.

ELIGIBILITY:
Inclusion Criteria:

* Impaired fasting glucose as defined by American Diabetes Association criteria: fasting plasma glucose level from 5.6 mmol/L (100 mg/dL) to 6.9 mmol/L (125 mg/dL)
* Body mass index (BMI) 25-34.9
* Age 18 and above• Weight stable: no more than 1 kg weight gain or loss during past 12 weeks

Exclusion Criteria:

* Fasting glucose >126 or <99 mg/dL
* BMI < 25 or >35
* Current/previous diagnosis of diabetes
* History of eating disorder or presence of active gastrointestinal disorders such as malabsorption syndromes
* Pregnancy or lactation Anemia, defined as hemoglobin level less than 10g/dl.
* Use of obesity pharmacotherapeutic agents within the last 6 months
* Use of over-the-counter anti-obesity agents (e.g. those containing phenylpropylamine , ephedrine and/or caffeine) within the last 3 months
* Chronic use of anti-inflammatory agents within the last four weeks
* Use of antioxidant supplements within the last four weeks including selenium, vitamin E, vitamin C and/or carotenoids
* Use of supplements containing any of the study compounds within the past four weeks
* Recent (current or past 12 weeks) use of any psychotropic medication
* Recent (past four weeks) initiation of or change in an exercise program
* Recent (past twelve weeks) initiation of hormone replacement therapy or change in HRT regimen
* Recent (past twelve weeks) initiation of hormonal birth control or change in hormonal birth control regimen
* Recent (past 12-weeks) history of tobacco use
* Any Condition that the P.I. considers adverse to the participant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Glucose Control | 28 days
  We will evaluate the effects of resveratrol/leucine and resveratrol/HMB for their ability to control glucose levels in persons without diabetes but with impaired fasting glucose

SECONDARY OUTCOMES:
Metabolic Markers | 28 days
  Secondary assessments will examine the effect of these nutritional supplements versus placebo on inflammation, fasting lipids, HbA1C, and fructosamine, longer term metabolic markers of risk in diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Niswender, MD,PHD, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Facility: Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Baur JA, Sinclair DA. Therapeutic potential of resveratrol: the in vivo evidence. Nat Rev Drug Discov. 2006 Jun;5(6):493-506. doi: 10.1038/nrd2060. Epub 2006 May 26. PMID 16732220
- [Background] Bordone L, Guarente L. Calorie restriction, SIRT1 and metabolism: understanding longevity. Nat Rev Mol Cell Biol. 2005 Apr;6(4):298-305. doi: 10.1038/nrm1616. PMID 15768047
- [Background] Verdin E, Hirschey MD, Finley LW, Haigis MC. Sirtuin regulation of mitochondria: energy production, apoptosis, and signaling. Trends Biochem Sci. 2010 Dec;35(12):669-75. doi: 10.1016/j.tibs.2010.07.003. Epub 2010 Sep 20. PMID 20863707
- [Background] Blum CA, Ellis JL, Loh C, Ng PY, Perni RB, Stein RL. SIRT1 modulation as a novel approach to the treatment of diseases of aging. J Med Chem. 2011 Jan 27;54(2):417-32. doi: 10.1021/jm100861p. Epub 2010 Nov 16. No abstract available. PMID 21080630
- [Background] Zemel MB. Role of calcium and dairy products in energy partitioning and weight management. Am J Clin Nutr. 2004 May;79(5):907S-912S. doi: 10.1093/ajcn/79.5.907S. PMID 15113738
- [Background] Zemel MB. Calcium and dairy modulation of obesity risk. Obes Res. 2005 Jan;13(1):192-3. doi: 10.1038/oby.2005.26. No abstract available. PMID 15761181
- [Background] Zemel MB, Sun X. Calcitriol and energy metabolism. Nutr Rev. 2008 Oct;66(10 Suppl 2):S139-46. doi: 10.1111/j.1753-4887.2008.00099.x. PMID 18844841
- [Background] Sun X, Zemel MB. Leucine and calcium regulate fat metabolism and energy partitioning in murine adipocytes and muscle cells. Lipids. 2007 Apr;42(4):297-305. doi: 10.1007/s11745-007-3029-5. Epub 2007 Feb 20. PMID 17406924